CLINICAL TRIAL: NCT04468594
Title: The Effect of Rigid Taping Versus Scapular Stabilizing Exercises on Pain and Function in Patients With Shoulder Subacromial Impingement Syndrome: a Randomized Controlled Trial
Brief Title: Rigid Taping Versus Scapular Stabilizing Exercises in Subacromial Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hail (Other)
Collaborators: Taif University (Other)
Responsible Party: Principal Investigator, Hisham Mohamed Hussein, Assistant Professor, University of Hail
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1234567890
Record Dates: First submitted 2020-07-03; First posted 2020-07-13 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Impingement Syndrome of Ankle
Keywords: Impingement Syndrome- rigid tape-scapular stabilizing
MeSH Terms: interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: double-blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: the process of allocation will be concealed using non transparent envelops that contain a code number. these codes indicated one of the three groups. the interpretation of these codes will be with an author who will not be involved in assessment or treatment procedures. At the day of the first intervention session, the code interpretation will be available
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rigid tape (Experimental): the rigid tapping technique using zinc oxide tape and protective tape (reference). With the participant assuming a relaxed standing position, the tape was applied bilaterally starting from the first to the last thoracic vertebra. A second tape was then applied to form a position of scapular depression and retraction. This tape was applied bilaterally and extended from the midpoint of the spine of the scapula to the last thoracic vertebra (figure ). This taping was applied for 12 weeks and changes every 3 days
  Interventions: Other: rigid tapping; Other: therapeutic exercises
- scapular stabilizing exercises (Experimental): scapular stabilizing exercises in the form of (1)wall slides with squat, (2) Wall push-ups with ipsilateral leg extension, (3) lawnmower with diagonal squat, (4) resisted retraction to scapula with opposite leg squat (5) robbery with squat. ten repetitions / exercises/ session were perform
  Interventions: Other: scapular stabilizing excercise; Other: therapeutic exercises
- control (Active Comparator): a standard physical therapy protocol will be introduced. This protocol consisted of (1) progressive strengthening exercises for rotator cuff muscles. The resistance was applied first by a red-colored elastic Thera-band. Then progressed, using the green-colored band. Each exercise was performed 10 times /session, (2) Self-stretching exercises for levator scapula, posterior deltoid, pectoralis minor, and latissimus dorsi muscles. Five repetitions of stretching were performed for each muscle per session
  Interventions: Other: therapeutic exercises

INTERVENTIONS:
Other: rigid tapping — Taping techniques We will use rigid tape and apply it bilaterally. In the rigid tape application, a combination pack of zinc oxide tape and the protective tape will be used. The protective tape will be applied first with no tension. To apply the rigid tape, subjects will be instructed to place their thoracic spine in a neutral position, the rigid tape will be applied bilaterally from the first to the twelfth thoracic vertebra. Subjects will be asked to retract and depress the scapula. The rigid tape will be applied diagonally from the middle of the scapular spine to the twelfth thoracic vertebra; this technique will be applied bilaterally. The rigid tape will be applied 3 times per week and will be applied for 6 weeks.
  Arms: rigid tape
Other: scapular stabilizing excercise — consisted of:
  1. wall slides with squat,
  2. wall push-ups plus ipsilateral leg extension,
  3. lawnmower with diagonal squat,
  4. resisted scapular retraction with contralateral leg squat and robbery with squat.
  5. Robbery with squat
  6. Resisted shoulder internal rotation with step
  7. Resisted shoulder external rotation with step
  8. Resisted full can with step All resisted exercises were performed with elastic bands with red color-coded resistance levels and progressed through green and blue bands The patient will perform 10 repetitions 3 sets to 15 repetitions 3 sets and 20 repetitions 3 sets weekly.
  Arms: scapular stabilizing exercises
Other: therapeutic exercises — 1. Pectoralis minor stretching
  2. Posterior shoulder stretching
  3. Levator scapula stretching
  4. Latissimus dorsi stretching ( stretching exercises will be 5 repetitions each session - 3 times per week)
  5. Resisted shoulder internal rotation
  6. Resisted shoulder external rotation
  7. Resisted full can (strengthening exercises will be 510 repetitions each session - 3 times per week) All resisted exercises were performed with elastic bands with red color-coded resistance levels and progressed through green and blue bands NOTE. All resisted exercises were progressed from starting 10 repetitions 3 sets to 15 repetitions 3 sets and 20 repetitions 3 sets weekly, supervising movement quality, presence of pain, and fatigue. If the subject achieves 20 repetitions 3 successfully, heavier resistance with resistance band color-coded loading prescribed from 10 repetitions 3 sets.

SUMMARY:
the current study tends to compare the effect of two different treatment techniques used in the rehabilitation of shoulder impingement syndrome. rigid tapping and scapular stabilizing exercises will be applied and the level of function and pain intensity will be measured before and after the intervention and at 3 months follow up. while both methods of treatment used previously, the comparison between their effects is not yet investigated and no data is available regarding the superiority of one over the other.

DETAILED DESCRIPTION:
Patients will be recruited through a verbal and written announcement from the customers of a local out-patient clinic. The appropriate number of patients, diagnosed with SIS, who will meet the inclusion criteria and accept to sign a consent form will join the study.

patients will be assigned randomly into three equal groups using permuted blocks of variable sizes. The first group rigid tape (RT) group will receive rigid taping plus a standard physical therapy protocol. The second group scapular stabilizing exercises (SSE) group will receive scapular stabilizing exercises plus the same standard protocol, and the third group (control group) will receive the standard protocol only.

The inclusion criteria were: positive 4 out of the following clinical signs: empty can test, Hawkins sign, Neer' sign, tenderness upon palpation of the greater tuberosity of the humerus, and painful movement between 60°_ and 120°(painful arc) Patients will be excluded if they demonstrate a previous history of shoulder surgery, cervical spine involvement, upper-limb fracture, adhesive capsulitis, joint instability, intraarticular corticosteroids injections within the last 2 months During the first interview, all patients will be checked for inclusion criteria. then undergo baseline assessment for pain level using a validated version of the Visual Analog Scale (VAS). Moreover, the functional level of the shoulder will be assessed using shoulder pain and disability index (SPADI). SPADI is a valid and reliable scale. it has a score ranging from 0 (normal) to 100 (complete disability). Pain and functional level will be assessed again after the end of the treatment period and after 3 months (following up) 12 weeks-rehabilitation program will be implemented for all patients with a frequency of 3 sessions/week. The RT group will receive a bilateral rigid taping technique using zinc oxide tape and along with the protective tape. With the participant assuming a relaxed standing position, the tape will be applied bilaterally starting from the first to the last thoracic vertebra. then, a second tape will be applied to the scapula while it assumes a position of scapular depression and retraction. This tape will be applied bilaterally and extended from the midpoint of the spine of the scapula to the last thoracic vertebra. This taping was applied for 12 weeks and changes every 2 days (3times per week) In addition to the rigid tape, a standard physical therapy protocol will be introduced. This standard protocol will consist of progressive strengthening exercises for rotator cuff muscles. The resistance will be applied first by a red-colored elastic Thera-band. Then progressed, using the green-colored band. Each exercise will be performed 10 times /session, Self-stretching exercises for levator scapula, posterior deltoid, pectoralis minor, and latissimus dorsi muscles. Five repetitions of stretching will be performed for each muscle per session In addition to the standard protocol, the SSE group will receive scapular stabilizing exercises in the form of wall slides with squat, Wall push-ups with ipsilateral leg extension, lawnmower with diagonal squat, resisted retraction to scapula with opposite leg squat robbery with squat. ten repetitions / exercises/ session were performed .

The CG will receive the standard protocol only Statistical analysis: SPSS (Version 16) for Windows will be used to analyze the obtained data. Mean± SD and percentage of differences will be calculated.

the current study tends to compare the effect of two different treatment techniques used in the rehabilitation of SIS. Rigid tapping and scapular stabilizing exercises will be applied then the level of function, and pain intensity will be measured before and after the intervention and at 3 months follow-up.

Detailed Description: Patients will be recruited through a verbal and written announcement from the customers of a local out-patient clinic. the appropriate sample size of patients diagnosed with SIS who will meet the inclusion criteria will join the study after signing the consent form.

patients will be assigned randomly into three equal groups using permuted blocks. The first group (RTG) received rigid taping plus a standard physical therapy protocol. The second group (SSEG) received scapular stabilizing exercises plus the same standard protocol, and the third group (control group) received the standard protocol only The inclusion criteria were: positive 4 out of the clinical signs: empty can test, Hawkins sign, Neer' sign, tenderness upon palpation of the greater tuberosity of the humerus, and painful movement between 60°_ and 120°(painful arc) Subjects will be excluded if they have a previous history of shoulder surgery, cervical spine involvement, upper-limb fracture, adhesive capsulitis, joint instability, intraarticular corticosteroids injections within the last 2 months During the first interview, all subjects will be checked for inclusion criteria. Eligible subjects will be assessed for pain level using a validated version of the Visual Analog Scale (VAS). Moreover, the functional level of the shoulder will be assessed using shoulder pain and disability index (SPADI). It is a valid and reliable scale with a score ranging from 0 (normal) to 100 (complete disability). Pain and functional level were assessed again after the end of the treatment period and after 3months (following up) 12 weeks-rehabilitation program will be implemented for all participants with a frequency of 3 sessions/week. The RT group will receive a bilateral rigid taping technique using zinc oxide tape and along with the protective tape. With the participant assuming a relaxed standing position, the tape will be applied bilaterally starting from the first to the last thoracic vertebra. then, a second tape will be applied to the scapulae while it assumes a position of scapular depression and retraction. This tape will be applied bilaterally and extended from the midpoint of the spine of the scapula to the last thoracic vertebra. This taping will be applied for 12 weeks and will be changed every 2 days (3times per week) In addition to the rigid tape, a standard physical therapy protocol will be conducted. This protocol will consist of progressive strengthening exercises for rotator cuff muscles. The resistance was applied first by a red-colored elastic Thera-band. Then progressed, using the green-colored band. Each exercise will be performed 10 times /session,( Self-stretching exercises for levator scapula, posterior deltoid, pectoralis minor, and latissimus dorsi muscles. Five repetitions of stretching will be performed for each muscle per session In addition to the standard protocol, the SSE group will receive scapular stabilizing exercises in the form of wall slides with squat, Wall push-ups with ipsilateral leg extension, lawnmower with diagonal squat, resisted retraction to scapula with opposite leg squat robbery with squat. ten repetitions / exercises/ session were performed .

The CG will receive the standard protocol only Statistical analysis: SPSS (Version 16) for Windows will be used to analyze the obtained data. Mean± SD and percentage of differences will be calculated.

ELIGIBILITY:
Inclusion Criteria:

Subjects having positive results to at least 4 of the following tests:

1. Neer impingement sign
2. Hawkins sign
3. pain during supraspinatus empty can test
4. the painful arc between 60⁰_ and 120⁰
5. tenderness when palpating the greater tuberosity of the humerus -

Exclusion Criteria:

Subjects will be excluded if they have;

* cervical spine involvement;
* the presence of a glenohumeral joint adhesive capsulitis, or instability;
* a history of previous shoulder surgery;
* upper-limb fracture;
* had systemic illnesses,
* receiving another physiotherapy treatment of this disorder in the past 6 weeks; or
* receiving steroid injection into or around the shoulder in the past 2 months.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
The Shoulder Pain and Disability Index (SPADI) | Change from Baseline Shoulder pain and function at 3 months"
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use. The SPADI takes 5 to 10 minutes for a patient to complete and is the only reliable and valid region-specific measure for the shoulder.

SECONDARY OUTCOMES:
pain (visual analouge scale) | Change from Baseline Shoulder pain at 3 months"
  scale with a score ranging from 0 (normal) to 100 (complete disability

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim M dewir, Assist .prof, Principal Investigator — physical therapy dep, College of Applied Medical Sciences, Taif University, S.A
Locations (1):
- University of Hail, Ha'il, Ha'il Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
this is the policy of the laboratory where the practical part will be conducted

REFERENCES:
- [Background] Buttagat V, Taepa N, Suwannived N, Rattanachan N. Effects of scapular stabilization exercise on pain related parameters in patients with scapulocostal syndrome: A randomized controlled trial. J Bodyw Mov Ther. 2016 Jan;20(1):115-122. doi: 10.1016/j.jbmt.2015.07.036. Epub 2015 Jul 26. PMID 26891646
- [Background] Cools AM, Witvrouw EE, Danneels LA, Cambier DC. Does taping influence electromyographic muscle activity in the scapular rotators in healthy shoulders? Man Ther. 2002 Aug;7(3):154-62. doi: 10.1054/math.2002.0464. PMID 12372312
- [Background] De Mey K, Danneels L, Cagnie B, Van den Bosch L, Flier J, Cools AM. Kinetic chain influences on upper and lower trapezius muscle activation during eight variations of a scapular retraction exercise in overhead athletes. J Sci Med Sport. 2013 Jan;16(1):65-70. doi: 10.1016/j.jsams.2012.04.008. Epub 2012 May 31. PMID 22658589
- [Background] Green S, Buchbinder R, Glazier R, Forbes A. Systematic review of randomised controlled trials of interventions for painful shoulder: selection criteria, outcome assessment, and efficacy. BMJ. 1998 Jan 31;316(7128):354-60. doi: 10.1136/bmj.316.7128.354. PMID 9487172
- [Background] Hebert LJ, Moffet H, McFadyen BJ, Dionne CE. Scapular behavior in shoulder impingement syndrome. Arch Phys Med Rehabil. 2002 Jan;83(1):60-9. doi: 10.1053/apmr.2002.27471. PMID 11782834
- [Background] Green S, Buchbinder R, Hetrick S. Physiotherapy interventions for shoulder pain. Cochrane Database Syst Rev. 2003;2003(2):CD004258. doi: 10.1002/14651858.CD004258. PMID 12804509
- [Background] Kalter J, Apeldoorn AT, Ostelo RW, Henschke N, Knol DL, van Tulder MW. Taping patients with clinical signs of subacromial impingement syndrome: the design of a randomized controlled trial. BMC Musculoskelet Disord. 2011 Aug 17;12:188. doi: 10.1186/1471-2474-12-188. PMID 21849055
- [Background] Kamkar A, Irrgang JJ, Whitney SL. Nonoperative management of secondary shoulder impingement syndrome. J Orthop Sports Phys Ther. 1993 May;17(5):212-24. doi: 10.2519/jospt.1993.17.5.212. PMID 8343779
- [Background] Kaya E, Zinnuroglu M, Tugcu I. Kinesio taping compared to physical therapy modalities for the treatment of shoulder impingement syndrome. Clin Rheumatol. 2011 Feb;30(2):201-7. doi: 10.1007/s10067-010-1475-6. Epub 2010 Apr 30. PMID 20443039
- [Background] Kibler WB, McMullen J, Uhl T. Shoulder rehabilitation strategies, guidelines, and practice. Orthop Clin North Am. 2001 Jul;32(3):527-38. doi: 10.1016/s0030-5898(05)70222-4. PMID 11888148
- [Background] Kuhn JE. Exercise in the treatment of rotator cuff impingement: a systematic review and a synthesized evidence-based rehabilitation protocol. J Shoulder Elbow Surg. 2009 Jan-Feb;18(1):138-60. doi: 10.1016/j.jse.2008.06.004. Epub 2008 Oct 2. PMID 18835532
- [Background] Lewis JS, Wright C, Green A. Subacromial impingement syndrome: the effect of changing posture on shoulder range of movement. J Orthop Sports Phys Ther. 2005 Feb;35(2):72-87. doi: 10.2519/jospt.2005.35.2.72. PMID 15773565
- [Background] Ludewig PM, Cook TM. Alterations in shoulder kinematics and associated muscle activity in people with symptoms of shoulder impingement. Phys Ther. 2000 Mar;80(3):276-91. PMID 10696154
- [Background] Ludewig PM, Reynolds JF. The association of scapular kinematics and glenohumeral joint pathologies. J Orthop Sports Phys Ther. 2009 Feb;39(2):90-104. doi: 10.2519/jospt.2009.2808. PMID 19194022
- [Background] McClure P, Greenberg E, Kareha S. Evaluation and management of scapular dysfunction. Sports Med Arthrosc Rev. 2012 Mar;20(1):39-48. doi: 10.1097/JSA.0b013e31824716a8. PMID 22311292
- [Background] McClure PW, Bialker J, Neff N, Williams G, Karduna A. Shoulder function and 3-dimensional kinematics in people with shoulder impingement syndrome before and after a 6-week exercise program. Phys Ther. 2004 Sep;84(9):832-48. PMID 15330696
- [Background] Miller P, Osmotherly P. Does scapula taping facilitate recovery for shoulder impingement symptoms? A pilot randomized controlled trial. J Man Manip Ther. 2009;17(1):E6-E13. doi: 10.1179/jmt.2009.17.1.6E. PMID 20046559